CLINICAL TRIAL: NCT06507111
Title: The Impact of Probiotic Supplementation on the Well-being of Women.
Brief Title: The Impact of Probiotics on Well-being in Women
Acronym: ProWOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cultech Ltd (Industry)
Collaborators: Comac Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ProWOME
Record Dates: First submitted 2024-07-03; First posted 2024-07-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Female; Healthy Aging
Keywords: Well-being; Probiotic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Lab4P Multi-strain Probiotic (comprising Lactobacilli and bifidobacteria species) with Vitamin C, Vitamin D and Zinc
  Interventions: Dietary Supplement: Lab4P
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lab4P — Lactobacillus acidophilus CUL-60, Lactobacillus acidophilus CUL-21, Lactobacillus plantarum CUL-66, Bifidobacterium bifidum CUL-20 and Bifidobacterium animalis subsp. lactis CUL-34 at a dose of 50 billion bacteria per/ day combined with vitamin C (80 mg/day), Vitamin D (400 IU/day) and Zinc (10 mg/day) on a microcrystaline cellulose (MCC) base
  Daily dose: 50 billion bacteria per day
  Arms: Active
Other: Placebo — MCC alone
  Arms: Placebo

SUMMARY:
An exploratory study to determine whether daily supplementation with a probiotic product impacts the overall well-being of women aged between 45 - 65

DETAILED DESCRIPTION:
It is generally accepted that there is a gradual decline in general well-being associated with aging. In previous studies with healthy adults receiving the Lab4P probiotic the outcomes indicated an overall improvement in general well-being and these findings provide the focus for the current trial which is investigating whether daily supplementation with the Lab4P probiotic product can impact upon the well-being of a cohort of women aged between 45 - 65 years (peri-menopausal/menopausal/post-menopausal).

The trial will be a double blinded, 2-arm, randomized, placebo-controlled, parallel group superiority study consisting of 50 women (gender as assigned at birth), aged between 45-65. The randomisation scheme will be generated by using a web-based interface using 1:1 allocation into 2 groups (block size 2).

The participants will make two site visits, the first visit for enrolment when they will be randomised, allocated their appropriate study product and their height, body weight and blood pressure will be measured. They will also be given a series of questionnaires assessing sleep (Athen Insomnia Scale), Mood (Hospital Anxiety and Depression Scale) and Quality of Life (Menopause Rating Scale) together with two cognitive tests (Word colour Stroop and Rey Auditory Verbal Learning Test (RAVLT)) to complete. A blood sample, a stool sample and a vaginal swab will be collected at this visit (if possible) and the participant will be given sample collection kits to take with them to collect futher samples prior to their second visit. They will be given a copy of each of the questionnaires and requested to be completed them and return by post at the study midpoint (day 56). They will also receive a copy of a Well-being diary that they will be asked to complete weekly throughout the study.

The second visit will take place at the end of the study (around day 112) and at that time the participants will bring the stool sample and vaginal swab collected at home and provide the final blood sample. At this time the participants will also complete each of the questionnaires (sleep, mood and quality of life) on site and repeat the Word Colour Stroop and RAVLT tests. The completed weekly Well-being diaries and any unused intervention will be returned. Scientists will use the information and samples collected to assess the benefits of taking the probiotic supplement.

It is considered that the daily intake of the probiotics will improve general wellbeing and mental health. Due to the chance that the use of the placebo, it is possible that any benefits will be confined to the participants who are randomly assigned the probiotic product. It is envisaged that the results generated from this study will enhance and improve our understanding of the benefits of daily probiotic supplementation.

There is no record of any adverse reactions associated with the regular consumption of this probiotic product but participants may experience mild side effects such as a change in bowel habit and/ or increased flatulence (intestinal gas) during the first few days of taking the supplement.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 45 to 65
2. Willing to provide faecal samples, blood samples and vaginal swabs
3. BMI of less than 30 kg/m2
4. Willing to maintain normal diet and lifestyle during the study
5. Willing to refrain from taking other probiotic supplements during the study
6. Normal (or corrected-to-normal) vision without colour blindness in order to complete the cognitive task

Exclusion Criteria:

1. No oral antibiotics within the last 3 months
2. No previous been involvement in a Cultech funded study
3. No regular consumption of probiotics within the last 1 month prior to the study
4. Premature menopause (onset before age of 40)
5. Given birth in the last 3 months, currently pregnant or planning pregnancy
6. Receiving hormone replacement therapy
7. Shift worker
8. Diagnosed with diabetes
9. Immunodeficient or undergoing immunosuppressive therapy
10. Diagnosed with arrhythmia, ventricular extrasystole or atrioventricular block
11. Diagnosed with a cardiovascular disease
12. Diagnosed with a severe systemic disease e.g. cancer, dementia, advanced organ failure.
13. Unexplained loss of weight in recent months

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Quality of Life Questionnaire | At Day 1, Day 56 and Day 112 ± 3 after trial start
  Quality of life questionnaire to evaluate the participants quality of life post probiotic supplementation. This QoL questionnaire uses a non-numeric, 5-point scale, ranking the presence and severity of symptoms as "none, mild, moderate, severe, and extremely severe".
Sleep Quality Questionnaire | At Day 1, Day 56 and Day 112 ± 3 after trial start
  Sleep quality questionnaire to measure the participants quality of sleep post probiotic supplementation. This sleep questionnaire uses the Athens Insomnia Scale and reports sleep quality using select phrases, and not a scored scale, such as "no problem, minor problem, considerable problems, serious problems". These phrases are question dependent.
Mood Questionnaire | At Day 1, Day 56 and Day 112 ± 3 after trial start
  Mood questionnaires to evaluate the participants mood post probiotic supplementation. This mood questionnaire is based off the Hospital Anxiety Depression Scale (HADS) and uses a four point scale for severity ranging from "0 - 3" with 0 being the lowest symptom severity and 3 being the highest symptom severity.

SECONDARY OUTCOMES:
Weekly Well-being Diary | Days 1, 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 77, 84, 91, 98, 105 and 112
  Weekly well-being diary to evaluate the participants general well-being post probiotic supplementation. This well-being diary records the frequency of days in the week that symptoms were experienced, this is between 1 - 7.
Bacterial composition of faecal samples via sequencing | At Day 1 and Day 112 ± 3 after trial start
  Shotgun metagenomic sequencing analysis to assess the bacterial composition of the faecal microbiome.
Bacterial composition of vaginal samples via sequencing | At Day 1 and Day 112 ± 3 after trial start
  Shotgun metagenomic sequencing analysis to assess the bacterial composition of the vaginal microbiome.
Blood plasma analysis for plasma lipids | At Day 1 and Day 112 ± 3 after trial start
  Blood plasma samples analysed for plasma lipids such as cholesterol and triglycerides.
Blood plasma analysis inflammatory markers | At Day 1 and Day 112 ± 3 after trial start
  Blood plasma samples analysed for plasma inflammatory markers such as IL-1B, TNFa, IL6, IL8, CCL2.

CONTACTS AND LOCATIONS:
Overall Officials: Daryn Michael, PhD, Principal Investigator — Cultech Ltd
Locations (1):
- Comac Medical, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol